CLINICAL TRIAL: NCT04480125
Title: The Efficacy and Safety of Azacitidine in Combination With Chidamide in the Treatment of Newly Diagnosed Peripheral T-Cell Lymphoma Unfit for Conventional Chemotherapy
Brief Title: Azacitidine Combined With Chidamide in the Treatment of Newly Diagnosed PTCL Unfit for Conventional Chemotherapy
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ruijin Hospital (Other)
Responsible Party: Principal Investigator, Zhao Weili, First Deputy Director，Hematology Department, Ruijin Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RJ-PTCL-2
Record Dates: First submitted 2020-07-19; First posted 2020-07-21 (Actual); Last update posted 2022-04-20 (Actual); Status verified 2022-04

CONDITIONS: Peripheral T-cell Lymphoma
Keywords: Peripheral T-cell lymphoma; Targeted therapy; Chemo-free therapy
MeSH Terms: conditions — Lymphoma, T-Cell, Peripheral | interventions — Azacitidine; N-(2-amino-5-fluorobenzyl)-4-(N-(pyridine-3-acrylyl)aminomethyl)benzamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Aza+Chida (Experimental): Azacitidine ivgtt D1-7 Chindamide 30mg,PO,twice a week Every 21 days for total 6 courses
  Interventions: Drug: Azacitidine; Drug: Chidamide

INTERVENTIONS:
Drug: Azacitidine — 100mg D1-7
Drug: Chidamide — 30mg BIW PO

SUMMARY:
This prospective, open-label, single-arm study will evaluate the efficacy and safety of azacitidine in combination with chidamide in treatment of newly diagnosed peripheral T-cell lymphoma unfit for conventional chemotherapy.

DETAILED DESCRIPTION:
Peripheral T-cell lymphoma (PTCL is a distinct and heterogeneous histopathologic subtype of non-Hodgkin lymphoma (NHL), accounting for ~10%. CHOP regimen has been widely used in PTCL patients even with unfavourable prognosis, with 5-year overall survival rate of 38.5%. Elderly patients seldom benefit from conventional CHOP regimen. A study showed that CR rate was only 18.1% in elderly patients (median age of 80 years old, ranging from 56 to 93 years old).

Azacitidine combined with romidepsin has been proved efficient in relasped or refractory PTCL, with CR rate of 55%. This prospective, open-label, single-arm study will evaluate the efficacy and safety of azacitidine in combination with Chidamide in treatment of newly diagnosed peripheral T-cell lymphoma unfit for conventional chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically confirmed peripheral T-cell lymphoma based on 2016 WHO classification
* Treatment naive
* Age ≥ 18 years
* Unfit for converntional chemotherapy meeting criteria as following but not limited to: age ≥75, ECOG >2，ADL<100 or CCI>1.
* Must has measurable lesion in CT or PET-CT prior to treatment
* Expected lifetime ≥ 3 months
* Informed consented

Exclusion Criteria:

* Has accepted localized or systemic anti-lymphoma treatment
* Has accepted autologous Stem cell transplantation before
* History of malignancy except for basal cell or squamous cell carcinoma of the skin or carcinoma in situ of the cervix prior to study treatment
* Uncontrollable cardio-cerebral vascular, coagulative, autoimmune, serious infectious disease
* Primary CNS lymphoma
* Left EF≤ 50%
* Lab at enrollment (Unless caused by lymphoma): Neutrophile<1.5*10^9/ L ;Platelet<75*10^9/L; ALT or AST >2*ULN; Creatinine>1.5*ULN
* Other uncontrollable medical condition that may that may interfere the participation of the study
* Not able to comply to the protocol for mental or other unknown reasons
* Patients with mentally disorders or other reasons unable to fully comply with the study protocol
* Pregnant or lactation
* HIV infection
* HBV-DNA and HCV-RNA undectable.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2020-06-20 (Actual); Primary Completion 2022-06-20 (Estimated); Study Completion 2024-06-20 (Estimated)

PRIMARY OUTCOMES:
Complete response rate | At the end of Cycle 6 (each cycle is 21 days)
  Percentage of participants with complete response was determined on the basis of investigator assessments according to 2014 Lugano criteria

SECONDARY OUTCOMES:
Overall response rate | At the end of Cycle 6 (each cycle is 21 days)
  Percentage of participants with overall response was determined on the basis of investigator assessments according to 2014 Lugano criteria
Progression free survival | Baseline up to data cut-off (up to approximately 4 years)
  Progression-free survival was defined as the time from the date of diagnosis until the date of the first documented day of disease progression or relapse, using 2014 Lugano criteria,or death from any cause, whichever occurred first.
Overall survival | Baseline up to data cut-off (up to approximately 4 years)
  Overall survival was defined as the time from the date of diagnosis to the date of death from any cause. Reported is the percentage of participants with event. of disease progression or relapse, using 2014 Lugano criteria,or death from any cause, whichever occurred first.
Duration of response | Baseline up to data cut-off (up to approximately 4 years)
  Time from first occurrence of documented CR or PR to disease progression/relapse, or death from any cause for participants with a response of CR or PR. Tumor assessments were performed with PET-CT.
Treatment related mortality | Baseline up to data cut-off (up to approximately 4 years)
  Percentage of death related with treatment on the basis of investigator assessments
Number of Participants With Treatment-Related Adverse Events as Assessed by CTCAE | Baseline up to data cut-off (up to approximately 4 years)
  An adverse event is any untoward medical occurrence in a participant administered a pharmaceutical product and which does not necessarily have to have a causal relationship with the treatment. An adverse event can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding, for example), symptom, or disease temporally associated with the use of a pharmaceutical product, whether or not considered related to the pharmaceutical product. Preexisting conditions which worsen during a study are also considered as adverse events
Change From Baseline in European Organization for Research and Treatment of Cancer Quality of Life Core 30 (EORTC QLQ-C30) Domain Scores | : Baseline (pre-dose [Hour 0] on Cycle1 Day1), Cycle3 Day 1, end of treatment (up to Month 6), every 3 months 1st year, every 6 months 2nd year, and 12 months thereafter up to data cut-off, up to approximately 4 years (cycle length = 21 days)
  The EORTC QLQ-C30 is a health-related quality of life questionnaire. A higher score indicates better quality of life, with changes of 5 to 10 points considered to be a minimally important difference to participants.

OTHER OUTCOMES:
Circulating free Deoxyribonucleic Acid (cfDNA) monitoring | Baseline up to data cut-off (up to approximately 4 years)
  CfDNA in peripheral blood assessed by local lab
Exploratory biomarker analysis | Baseline up to data cut-off (up to approximately 4 years)
  Exploratory biomarker to predict treatment response and survival

CONTACTS AND LOCATIONS:
Overall Officials: Weili Zhao, Study Chair — Ruijin Hospital
Locations (1):
- Shanghai Ruijin Hospital, Shanghai, China